CLINICAL TRIAL: NCT05649436
Title: Assessment of Developmental Status and Locomotor Balance in Healthy Children. A Normative Study.
Brief Title: Assessment of Developmental Status and Locomotor Balance in Healthy Children.
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/22/00736 Duaa Ijaz
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Development, Child
Keywords: balance; developmental milestone; locomotor balance; proprioception; ages and stages questionnaire; timed up and go test

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess developmental milestones and balance in children in Pakistan. We are using Ages and Stages Questionnaire for developmental milestones and Timed up and Go test for balance.

DETAILED DESCRIPTION:
We will visit daycare centers and primary schools to collect data and compare them to cut off values provided in the scale. After scoring each domain, scores will tell whether child needs further investigation or he is healthy.

ELIGIBILITY:
Inclusion Criteria:

* 2 months to 5 years of age
* Families living in urban areas
* Families with financial stability when the child was growing

Exclusion Criteria:

* Multiple Pregnancies of mother
* A known history of diabetes of mother
* Uneducated Mother
* A known history of psychological problems of parents
* Impaired Cognition of Children
* Deafness or Blindness of Children
* Children with 36 weeks or less gestational periods

Ages: 2 Months to 5 Years | Sex: All
Age Groups: Child
Study Population: daycare centers primary schools
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Ages and Stages Questionnaire | last one week
  It is parent-completed questionnaires for young children. It ranges from age 1 to 60 months and consists of 19 different questionnaires.The questionnaires cover over five different domains: communication, gross motor, fine motor, problem solving and personal social skills.If the child scores below cut off value he needs further medical assessment otherwise he is healthy. Cut off values are different for each domain.
Timed Up and Go test | last one week
  Begin by having the patient sit back in a standard arm chair and identify a line 3 meters, or 10 feet away, on the floor. 2 On the word "Go," begin timing. 3 Stop timing after patient sits back down. 4 Record time. Observe the patient's postural stability, gait, stride length, and sway.

CONTACTS AND LOCATIONS:
Overall Officials: shabana ashraf, Phd, Principal Investigator — Riphah International University
Locations (1):
- Govt College of Technology for women, Day care center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fauls JR, Thompson BL, Johnston LM. Validity of the Ages and Stages Questionnaire to identify young children with gross motor difficulties who require physiotherapy assessment. Dev Med Child Neurol. 2020 Jul;62(7):837-844. doi: 10.1111/dmcn.14480. Epub 2020 Feb 11. PMID 32043571
- [Background] Agarwal PK, Shi L, Daniel LM, Yang PH, Khoo PC, Quek BH, Zheng Q, Rajadurai VS. Prospective evaluation of the Ages and Stages Questionnaire 3rd Edition in very-low-birthweight infants. Dev Med Child Neurol. 2017 May;59(5):484-489. doi: 10.1111/dmcn.13307. Epub 2016 Nov 24. PMID 27882544
- [Background] Park JH, Hwangbo G. The effect of trunk stabilization exercises using a sling on the balance of patients with hemiplegia. J Phys Ther Sci. 2014 Feb;26(2):219-21. doi: 10.1589/jpts.26.219. Epub 2014 Feb 28. PMID 24648635
- [Background] Verbecque E, Vereeck L, Boudewyns A, Van de Heyning P, Hallemans A. A Modified Version of the Timed Up and Go Test for Children Who Are Preschoolers. Pediatr Phys Ther. 2016 winter;28(4):409-15. doi: 10.1097/PEP.0000000000000293. PMID 27661232
- [Background] Villar J, Fernandes M, Purwar M, Staines-Urias E, Di Nicola P, Cheikh Ismail L, Ochieng R, Barros F, Albernaz E, Victora C, Kunnawar N, Temple S, Giuliani F, Sandells T, Carvalho M, Ohuma E, Jaffer Y, Noble A, Gravett M, Pang R, Lambert A, Bertino E, Papageorghiou A, Garza C, Stein A, Bhutta Z, Kennedy S. Neurodevelopmental milestones and associated behaviours are similar among healthy children across diverse geographical locations. Nat Commun. 2019 Jan 30;10(1):511. doi: 10.1038/s41467-018-07983-4. PMID 30700709
- [Background] Osoba MY, Rao AK, Agrawal SK, Lalwani AK. Balance and gait in the elderly: A contemporary review. Laryngoscope Investig Otolaryngol. 2019 Feb 4;4(1):143-153. doi: 10.1002/lio2.252. eCollection 2019 Feb. PMID 30828632